CLINICAL TRIAL: NCT06214871
Title: A Prospective Study To Evaluate Safety and Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) For Neuroenhancement
Brief Title: rTMS for Neuroenhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gerrish MedEsthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-001
Record Dates: First submitted 2023-12-06; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Transcranial Magnetic Stimulation

SUMMARY:
The purpose of this pilot study is to evaluate the effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Sleep Quality, Mood and Memory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 22 to 70 years of age
* Freely provides written informed consent
* In good general health, as ascertained by medical history
* If female, not breastfeeding, no known or suspected pregnancy, a status of non- childbearing potential or use of an acceptable form of birth control
* If subject is in menopausal transition, the subject must be stabilized on hormonal treatment.
* Subject scored a 2 or higher on PHQ-9 sleep related question (#3), OR subject scored 2 or more on at least 2 QIDS-SR sleep related questions (#'s 1-4)
* If subject is on any psychiatric or sleep medication, dose must be stable for two weeks prior to enrollment and remain stable throughout the trial.

Exclusion Criteria:

* Subject satisfies any one or more of the contraindications for TMS Therapy per current treatment guidelines as determined by the PI.
* History of head trauma associated with loss of consciousness or diagnosed as concussion.
* History of fainting, syncope, hearing problems or ringing in the ears (tinnitus)
* Has any metallic implant(s) in or near the head (e.g., pacemaker, defibrillator, neurostimulator, etc.) including any splinters, fragments, clips, etc.
* Has an implanted stimulator device (including device leads) in or near the head.

  (e.g. deep brain stimulator, cochlear implant, vagus nerve stimulator.)
* Has medication infusion device.
* Subjects with any prior TMS or MRI complications which, in the opinion of the investigator, might interfere with safety, study participation, or which might confound data interpretation,
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR), with the exception of nicotine dependence.
* Current diagnosis or known history of neurologic or neuropsychiatric disease (e.g., epilepsy, convulsion, seizure)
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent with study participation.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality - Jenkins Sleep Scale | Various - Over 8 weeks
  Jenkins Sleep Scale (Score can be from 0-20; higher scores equal lesser sleep quality)
Sleep Quality - PHQ-9 (Patient Health Questionnaire-9) | Various - Over 8 Weeks
  PHQ-9 (Question #3 score can be 0-3; higher score equal lesser sleep quality)
Sleep Quality - QIDS-SR (Quick Inventory of Depressive Symptomatology - Self Report) | Various - Over 8 Weeks
  QIDS-SR (Questions #1-#4 each question can be 0-3; higher score equals lesser sleep quality)

SECONDARY OUTCOMES:
Mood - PANAS (Positive and Negative Affect Schedule) | Various - Over 8 weeks
  Assessments; PANAS (20 Questions; The total score is calculated by finding the sum of the 10 positive items, and then the 10 negative items. Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect)
Memory - RAVLT Immediate Recall (Rey Auditory Verbal Learning Test) | Various - Over 8 weeks
  Assessment; RAVLT Immediate (the sum of scores from 5 first trials (Trials 1 to 5)),
Mood - SAMMS (Sleep, Anxiety, Mood, Memory Survey) | Various - Over 8 Weeks
  SAMMS (8 Questions; Total score ranges from 0-80; 2 of the questions are related to Mood and a higher score is better mood)
Mood - VAMS (Visual Analog Mood Scale) | Various - Over 8 Weeks
  VAMS (7 Questions; Total score can range from 0-70; higher scores represent better Mood)
Memory - RAVLT Delayed Recall | Various - Over 8 weeks
  RAVLT Forgetting (the score of Trial 5 minus score of the delayed recall)

CONTACTS AND LOCATIONS:
Locations (1):
- Gerrish MedEsthetics, Vienna, Virginia, United States